CLINICAL TRIAL: NCT04412668
Title: A Randomized Double-Blind Placebo-Controlled Study to Evaluate the Safety and Efficacy of ATYR1923 In Adult Patients With Severe Pneumonia Related to SARS-CoV-2 Infection (COVID-19)
Brief Title: Study to Evaluate the Safety and Efficacy of ATYR1923 (Efzofitimod) In Participants With Severe Pneumonia Related to COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATYR1923-C-003
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2 (COVID-19) Severe Pneumonia
Keywords: SARS-CoV-2; CoV-2; ATYR1923 (efzofitimod); acute respiratory distress syndrome; ARDS; SARS-CoV-2 Infection; COVID-19; Severe Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to a single intravenous (IV) dose of efzofitimod 1 mg/kg, efzofitimod 3 mg/kg, or placebo matched to efzofitimod.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigator, Sponsor, and participant will be blinded to treatment assignment; study center pharmacy personnel will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efzofitimod 1 mg/kg (Experimental): Participants will receive single dose of efzofitimod 1 milligrams/kilograms (mg/kg) IV infusion on Day 1.
  Interventions: Drug: Efzofitimod 1 mg/kg
- Efzofitimod 3 mg/kg (Experimental): Participants will receive single dose of efzofitimod 3 mg/kg IV infusion on Day 1.
  Interventions: Drug: Efzofitimod 3 mg/kg
- Placebo (Placebo Comparator): Participants will receive placebo matched to efzofitimod IV infusion on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efzofitimod 1 mg/kg — Concentrate for solution for infusion
  Arms: Efzofitimod 1 mg/kg
Drug: Efzofitimod 3 mg/kg — Concentrate for solution for infusion
  Arms: Efzofitimod 3 mg/kg
Drug: Placebo — Concentrate for solution for infusion
  Arms: Placebo

SUMMARY:
To evaluate the safety and preliminary efficacy of efzofitimod, compared to placebo matched to efzofitimod, in hospitalized participants with SARS-CoV-2 (COVID-19) severe pneumonia not requiring mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of SARS-CoV-2 infection by polymerase chain reaction (PCR).
* Severe pneumonia related to SARS-CoV-2 infection, defined as fever or suspected respiratory infection with radiographic abnormalities suggestive of viral pneumonia, plus at least 1 of the following:

  * Respiratory rate >30 breaths/minute;
  * Severe respiratory distress, as determined by the Investigator;
  * Oxygen saturation (SpO2) ≤93% on room air.

Exclusion Criteria:

* Participant is intubated/mechanically ventilated.
* In the opinion of the Investigator, participant's progression to death is imminent.
* Treatment with immunosuppressant/immunotherapy drugs, including but not limited to interleukin (IL)-6 inhibitors, tumor necrosis factor-alpha (TNF-α) inhibitors, anti-IL-1 agents and janus kinase inhibitors within 5 half-lives or 30 days prior to Day 1.
* Use of chronic (>30 days) oral corticosteroids for a non-COVID-19-related condition in a dose higher than prednisone 10 mg or equivalent per day.
* Weight >165 kg or <40 kg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - aTyr Investigative Site, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Anne Arundel Medical Center, Annapolis, Maryland
  - aTyr Investigative Site, Vineland, New Jersey
  - aTyr Investigative Site, Toledo, Ohio
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- Puerto Rico (2):
  - Alliance Medical Service, Cardio Pulmonary Research, Guaynabo
  - Manati Medical Center, Manatí

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Efzofitimod 1 mg/kg: Participants received single dose of efzofitimod 1 milligrams/kilograms (mg/kg) intravenous (IV) infusion on Day 1.
- Efzofitimod 3 mg/kg: Participants received single dose of efzofitimod 3 mg/kg IV infusion on Day 1.
- Placebo: Participants received placebo matched to efzofitimod IV infusion on Day 1.
Period: Overall Study
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Started | 14 | 12 | 10
Received at Least 1 Dose of Study Drug | 10 | 12 | 10
Completed | 7 | 12 | 10
Not Completed | 7 | 0 | 0
Not completed — Death - multiple comorbidities | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Other than Specified | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set was defined as all randomized participants who received any amount of study drug. Participants were summarized and analyzed 'as treated' (that is, by actual treatment group).
Groups:
- Efzofitimod 1 mg/kg: Participants received single dose of efzofitimod 1 mg/kg IV infusion on Day 1.
- Total: Total of all reporting groups
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo | Total
Number analyzed (Participants) | 10 | 12 | 10 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.08) | 56.5 (11.41) | 52.8 (10.51) | 55.2 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 14
  Male | 5 | 6 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 7 | 17
  Not Hispanic or Latino | 6 | 5 | 3 | 14
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 6 | 4 | 3 | 13
  More than one race | 2 | 5 | 3 | 10
  Unknown or Not Reported | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. AEs were defined as any untoward medical occurrence in a participant administered study drug and that does not necessarily have a causal relationship with the study drug. Worsening of a pre-existing medical condition should have been considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. SAEs were defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 60
Population: Safety Set was included all randomized participants who received any amount of study drug. Participants were summarized and analyzed 'as treated' (that is, by actual treatment group).
Measure: Count of Participants; unit: Participants
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 10 | 12 | 10
Participants
  TEAEs | 8 | 7 | 7
  SAEs | 5 | 0 | 0

2. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge was based on Kaplan-Meier estimate and was calculated as: discharge date - study drug administration date. Participants who died during hospitalization were censored at death date. Participants who remained hospitalized at end of study (EOS) were censored at EOS visit.
Time Frame: Baseline up to Day 60
Population: Modified intention-to-treat set (mITT Set) included all participants randomized who had received any amount of study drug. Participants were summarized and analyzed 'as randomized' (that is, by randomized treatment group).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 10 | 12 | 10
days | 7.0 [3.0 to 31.0] | 5.5 [2.0 to 6.0] | 4.5 [1.0 to 7.0]

3. Secondary Outcome: Time to Recovery (World Health Organization [WHO] Ordinal Scale Score ≤3)
Description: Time to recovery was based on Kaplan-Meier estimate and was calculated as: date of first time with a WHO scale score ≤3 - study drug administration date or date of discharge from hospital - study drug administration date, whichever occurred first. In the case that a participant did not reach WHO scale score ≤3 criteria, the participant was censored at EOS visit.
Time Frame: Baseline up to Day 60
Population: mITT set included all participants randomized who had received any amount of study drug. Participants were summarized and analyzed 'as randomized' (that is, by randomized treatment group).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 10 | 12 | 10
days | 7.0 [2.0 to 31.0] | 5.5 [2.0 to 6.0] | 4.5 [1.0 to 7.0]

4. Secondary Outcome: Number of Participants Who Achieved Recovery (WHO Ordinal Scale Score ≤3) by Day 14 and Day 28
Description: The number of participants was the non-missing value at the visit, which was used as the denominator for percentage calculation.
Time Frame: Baseline through Day 14 and Day 28
Population: mITT set included all participants randomized who had received any amount of study drug. Participants were summarized and analyzed 'as randomized' (that is, by randomized treatment group). Here, Number of Participants Analyzed signifies those who were evaluable for this outcome measure and Number Analyzed signifies those who were evaluable at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 6 | 12 | 10
Participants
  Day 14: number analyzed (Participants) | 5 | 10 | 8
  Day 14 | 4 | 9 | 7
  Day 28 | 5 | 11 | 9

5. Secondary Outcome: Number of Days With Supplemental Oxygen (O2)
Description: Number of days with supplemental O2 was calculated as stop date of supplemental O2 - start date of supplemental oxygen +1, if supplemental O2 started after study drug administration; otherwise, number of days with supplemental O2 was calculated as stop date of supplemental O2 - date of study drug administration +1. If there were multiple periods of supplemental O2, total days were the sum of each period.
Time Frame: Baseline up to Day 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 10 | 12 | 10
days | 10.4 (17.65) | 13.7 (16.05) | 10.1 (15.72)

6. Secondary Outcome: Number of Days With Fever (Temperature >100.4ºF [38.0ºC])
Description: Number of days with fever was calculated as stop date of fever - start date of fever +1, if fever started after study drug administration; otherwise, number of days with fever was calculated as stop date of fever - date of study drug administration +1. If there were multiple periods of fever, total days was the sum of each period.
Time Frame: Baseline up to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 10 | 12 | 10
days | 0.1 (0.32) | 0.1 (0.29) | 0.0 (0.00)

7. Secondary Outcome: Number of Participants With a Change From Baseline in World Health Organization (WHO) Ordinal Scale Score on Day 60
Description: WHO ordinal scale rated the clinical improvement of the participants on a scale of 0-8, where 0=No clinical or virological evidence of infection, 1=No limitation of activities, 2=limitation of activities, 3=Hospitalized, no oxygen therapy, 4=Oxygen by mask or nasal prongs, 5=Non-invasive ventilation or high flow oxygen, 6=Intubation and mechanical ventilation, 7=Ventilation + additional organ support, 8=Death. Change from Baseline data were represented on a scale of -7 to 4, where -7=a better change from Baseline score and 4=a worse change from Baseline score. Change from Baseline was derived as: visit value - Baseline value.
Time Frame: Baseline, Day 60
Population: mITT set included all participants randomized who had received any amount of study drug. Participants were summarized and analyzed 'as randomized' (that is, by randomized treatment group). Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 6 | 12 | 10
Participants
  -7 | 0 | 0 | 0
  -6 | 0 | 0 | 0
  -5 | 0 | 0 | 1
  -4 | 2 | 8 | 4
  -3 | 3 | 4 | 4
  -2 | 1 | 0 | 1
  -1 | 0 | 0 | 0
  0 | 0 | 0 | 0
  1 | 0 | 0 | 0
  2 | 0 | 0 | 0
  3 | 0 | 0 | 0
  4 | 0 | 0 | 0

8. Secondary Outcome: Time to Improvement From Inpatient Hospital Admission Based on at Least a 1-Point Reduction in WHO Ordinal Scale Score
Description: Time to improvement was based on Kaplan-Meier estimate and was defined as the date of decrease in WHO scale compared to Baseline by at least 1 point - study drug administration date or date of discharge from hospital - study drug administration date, whichever occurred first. In the case that a participant did not reach an improvement, the participant was censored at end of study date.
Time Frame: Baseline up to Day 60
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
Number analyzed (Participants) | 10 | 12 | 10
days | 5.0 [1.0 to 10.0] | 4.0 [2.0 to 6.0] | 3.0 [1.0 to 5.0]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 60
Description: Safety Set was defined as all randomized participants who received any amount of study drug. Participants were summarized and analyzed 'as treated' (that is, by actual treatment group).
Arm/Group | Efzofitimod 1 mg/kg | Efzofitimod 3 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/10 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/10 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 7/12 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efzofitimod 1 mg/kg (N=10) | Efzofitimod 3 mg/kg (N=12) | Placebo (N=10)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efzofitimod 1 mg/kg (N=10) | Efzofitimod 3 mg/kg (N=12) | Placebo (N=10)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood chloride decreased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Carbon dioxide increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0
Hepatitis B virus test positive (Investigations) | 1 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 1
Prothrombin time ratio increased (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Genital candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT04412668/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT04412668/SAP_001.pdf